CLINICAL TRIAL: NCT00707746
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess Safety and Efficacy of ISIS 301012 Administration in High Risk Statin Intolerant Subjects
Brief Title: Safety and Efficacy Study of ISIS 301012 (Mipomersen) Administration in High Risk Statin Intolerant Subjects
Acronym: ASSIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301012-CS19; 2007-005140-24 (EudraCT Number)
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Results first posted 2013-04-05 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Metabolic Diseases; Hyperlipidemias; Metabolic Disorder; Hypercholesterolemia; Dyslipidemias; Lipid Metabolism Disorders
Keywords: statin intolerant; hypercholesterolemia
MeSH Terms: conditions — Metabolic Diseases; Hyperlipidemias; Hypercholesterolemia; Dyslipidemias; Lipid Metabolism Disorders | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 1 mL placebo saline, weekly subcutaneous injections for 26 weeks
  Interventions: Drug: placebo
- Mipomersen (Experimental): 200 mg (1 mL), weekly subcutaneous injections for 26 weeks
  Interventions: Drug: mipomersen

INTERVENTIONS:
Drug: mipomersen
  Other Names: ISIS 301012; mipomersen sodium; Kynamro™
  Arms: Mipomersen
Drug: placebo
  Other Names: placebo saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine safety and efficacy of mipomersen (ISIS 301012) in the reduction of total cholesterol, low density lipoprotein cholesterol (LDL-C), and apolipoprotein B (apoB) in high risk subjects intolerant to statins.

DETAILED DESCRIPTION:
In humans, apoB is the principal apolipoprotein of the atherogenic lipoproteins, comprising very low-density lipoprotein (VLDL), intermediate density lipoprotein (IDL) and low density lipoprotein (LDL). ApoB messenger ribonucleic acid (mRNA) is abundantly present in the liver. Within the endoplasmatic reticulum, apoB requires lipidation by microsomal triglyceride transfer protein, which allows apoB to be incorporated in the VLDL particle within the lumen of the endoplasmatic reticulum. Non-lipidated apoB is readily degraded via ubiquitination. Notably, apoB within the VLDL particle is obligatory for hepatic secretion of VLDL. ApoB remains present within the VLDL-metabolism pathway, from secretion to clearance of the end product LDL by the liver LDL receptor. As a consequence, apoB reliably reflects the total burden of atherogenic lipoproteins. Thus, apoB carries strong prognostic value for cardiovascular events, which exceeds the predictive value of LDL-C. Conversely, decreased levels of apoB (e.g. in familial hypobetalipoproteinemia) have been associated with reduced levels of atherosclerosis. These genetic observations have prompted interest in pharmacologic inhibition of apoB synthesis.

Mipomersen (ISIS 301012) is an antisense drug targeted to human apoB, the principal apolipoprotein of LDL and its metabolic precursor, VLDL. Mipomersen (ISIS 301012) is complementary to the coding region of the mRNA for apoB, binding by Watson and Crick base pairing. The hybridization (binding) of mipomersen (ISIS 301012) to the cognate mRNA results in Ribonuclease (RNase) H-mediated degradation of the cognate mRNA, thus inhibiting translation of the apoB protein.

This was a randomized, double-blind, placebo-controlled Phase 2 study to assess the safety and efficacy of mipomersen administration in high-risk statin-intolerant patients with hypercholesterolemia. This study consisted of a ≤3-week screening period, 26 weeks of treatment, and a 24-week post-treatment follow-up period.

Eligible patients were randomized in a 2:1 ratio to receive mipomersen 200 mg or matching volume placebo subcutaneous (SC) injections weekly.

Following the screening visit, eligible patients returned to the study center for clinical evaluation every week for study drug administration and assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of statin intolerance
* Diagnosis of Coronary Artery Disease (CAD)
* Diagnosis of hypercholesterolemia
* Stable weight for > 6 weeks

Exclusion Criteria:

* Significant health problems in the recent past (≤24 weeks) including heart attack, heart surgery, heart failure, uncontrolled hypothyroidism, blood disorders, digestive problems, disease of central nervous system, cancer, liver or renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Amsterdam, Netherlands

REFERENCES:
- [Derived] Visser ME, Wagener G, Baker BF, Geary RS, Donovan JM, Beuers UH, Nederveen AJ, Verheij J, Trip MD, Basart DC, Kastelein JJ, Stroes ES. Mipomersen, an apolipoprotein B synthesis inhibitor, lowers low-density lipoprotein cholesterol in high-risk statin-intolerant patients: a randomized, double-blind, placebo-controlled trial. Eur Heart J. 2012 May;33(9):1142-9. doi: 10.1093/eurheartj/ehs023. Epub 2012 Apr 16. PMID 22507979
- [Derived] Patel N, Hegele RA. Mipomersen as a potential adjunctive therapy for hypercholesterolemia. Expert Opin Pharmacother. 2010 Oct;11(15):2569-72. doi: 10.1517/14656566.2010.512006. PMID 20707601

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 42 patients were screened, 34 participants were randomized, and 33 participants were treated: 21 participants to mipomersen and 12 participants to placebo.
Groups:
- Mipomersen: 200 mg (1 mL) of mipomersen, weekly subcutaneous injections for 26 weeks
Period: Treatment Period
Arm/Group | Placebo | Mipomersen
Started | 12 | 22
Full Analysis Set (FAS) and Safety Set | 12 (FAS: Treated patients with a valid baseline & post-baseline LDL-C measurement) | 21 (FAS: Treated patients with a valid baseline & post-baseline LDL-C measurement)
Completed | 10 | 17
Not Completed | 2 | 5
Not completed — Adverse Event | 2 | 4
Not completed — Ineligibility | 0 | 1
Period: Follow-up Period
Arm/Group | Placebo | Mipomersen
Started | 12 | 21
Completed | 12 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mipomersen | Total
Number analyzed (Participants) | 12 | 21 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (8.7) | 55.6 (6.8) | 54.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 4 | 11 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 21 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 20 | 32
  Black | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.06 (2.49) | 26.46 (3.25) | 26.31 (2.96)
Waist/hip Ratio [Mean (Standard Deviation); unit: ratio] | 0.92 (0.09) | 0.93 (0.08) | 0.93 (0.08)
Metabolic syndrome [Number; unit: participants] — A participant was classified as having metabolic syndrome if any 3 of the following risk factors existed: 1) Waist circumference ≥102 cm (men) or ≥88 cm (women); 2) Triglycerides ≥150 mg/dl *; 3) High density lipoprotein cholesterol <40 mg/dl (men) or <50 mg/dl (women)*; 4) Systolic blood pressure ≥130 or diastolic ≥85 mmHg *; 5) Fasting glucose ≥100 mg/dl *.
  * = or on medication for the specified risk factor.
  participants
    No | 4 | 12 | 16
    Yes | 8 | 9 | 17
Tobacco Use [Number; unit: participants]
  Current | 2 | 6 | 8
  Non-current | 5 | 9 | 14
  Never | 5 | 6 | 11
Alcohol use [Number; unit: participants]
  Current | 8 | 16 | 24
  Non-current | 2 | 3 | 5
  Never | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at the Primary Efficacy Time Point
Description: LDL-C was measured in mg/dL. Samples were taken following an overnight fast. For patients with triglycerides <400 mg/dL, LDL-C was obtained using Friedewald's calculation; and for patients with triglycerides ≥400 mg/dL, LDL-C was directly measured by the central laboratory using ultracentrifugation. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: Baseline (the average of the screening and Day 1 pre-treatment assessments) and the Primary Efficacy Time point (PET; Week 28 or the post-baseline visit closest to 14 days after the last dose).
Population: The Full Analysis Set, which consisted of all randomized patients who received at least 1 injection of study drug (mipomersen or placebo) and with a valid baseline and at least 1 post-baseline LDL-C measurement.
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | -2.0 (8.40) | -47.3 (18.43)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; It was estimated that the standard deviation of the percent change in LDL-C was 20%. A sample size of 30 patients was planned for this study: 20 patients in the mipomersen group and 10 patients in the placebo group. A 2-sided t-test with an alpha level of 0.05 was expected to provide ≥90% power to detect a 30% difference in LDL-C percent reduction between the 2 groups (35% reduction for the mipomersen group and 5% reduction for the placebo group); Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance was concluded if p ≤ 0.05

2. Primary Outcome: Low-density Lipoprotein Cholesterol at Baseline and the Primary Efficacy Time Point
Description: The primary efficacy time point (PET) was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 243.7 (65.6) | 241.9 (90.8)
  Primary efficacy time point | 236.3 (52.8) | 128.3 (74.2)

3. Primary Outcome: Summary of Participants With Adverse Events
Description: The on-treatment time frame spanned the time during which the study drug was administered until the later of the primary efficacy time point and 14 days beyond the last study drug date.
  Adverse events (AEs) were considered related if assessed by the Investigator as possibly, probably or definitely related to study drug.
  Severity was assessed as:
  * Mild-symptom barely noticeable to the patient or do not make the patient uncomfortable;
  * Moderate-symptom makes the patient uncomfortable, affects performance of daily activities;
  * Severe-symptom causes the patient severe discomfort, may cause cessation of treatment with the study drug.
  Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention.
Time Frame: Pre-treatment (prior to first dose), On-treatment (Day 1 to week 28), Post-treatment (Week 28-52)
Population: Safety set of all randomized participants who received at least one injection of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
participants
  Pre-treatment adverse events (AEs) | 3 | 7
  Post-treatment AEs | 9 | 20
  On-treatment AEs | 12 | 21
  On-treatment AEs-related | 12 | 21
  On-treatment AEs-mild | 6 | 5
  On-treatment AEs-moderate | 5 | 16
  On-treatment AEs-severe | 1 | 0
  On-treatment AEs-leading to trt discontinuation | 2 | 4
  On-treatment Serious Adverse Events (SAEs) | 1 | 0
  On-treatment SAEs-related | 1 | 0
  On-treatment SAEs-mild | 0 | 0
  On-treatment SAEs-moderate | 0 | 0
  On-treatment SAEs-severe | 1 | 0
  On-treatment SAEs-leading to trt discontinuation | 1 | 0
  Deaths | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Primary Efficacy Time Point
Description: Apolipoprotein B was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | -4.0 (8.40) [-8.8 to 0.5] | -45.8 (18.43) [-57.5 to -34.4]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank sum — Inflation of type 1 error was controlled by specifying a small number of secondary parameters and a sequential inferential approach in which inferential conclusions about each successive parameter required statistical significance of the prior one

5. Secondary Outcome: Apolipoprotein B at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 180 (65.6) [145 to 196] | 177 (90.8) [142 to 205]
  Primary efficacy time point | 173 (52.8) [143 to 187] | 96 (74.2) [66 to 110]

6. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at the Primary Efficacy Time Point
Description: Total cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | -1.7 (6.46) [-8.8 to 0.5] | -36.9 (14.66) [-57.5 to -34.4]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]

7. Secondary Outcome: Total Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 322.3 (66.2) | 318.9 (91.8)
  Primary efficacy time point | 314.5 (53.0) | 200.1 (77.6)

8. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: Non-high-density lipoprotein cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | -1.9 (7.06) [-8.8 to 0.5] | -45.6 (18.22) [-57.5 to -34.4]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]

9. Secondary Outcome: Non-High-Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 273.5 (65.3) | 270.1 (92.9)
  Primary efficacy time point | 266.0 (53.0) | 147.7 (81.1)

10. Other Pre Specified Outcome: Percent Change From Baseline in Triglycerides at the Primary Efficacy Time Point
Description: Triglycerides were measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | 5.0 (26.81) | -27.0 (30.21)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.005, t-test, 2 sided — Statistical significance was concluded if p ≤0.05. No further adjustments were made for tertiary parameters

11. Other Pre Specified Outcome: Triglycerides at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 149.0 (63.9) | 141.4 (50.9)
  Primary efficacy time point | 149.3 (62.4) | 97.3 (47.3)

12. Other Pre Specified Outcome: Percent Change From Baseline in Lipoprotein (a) at the Primary Efficacy Time Point
Description: Lipoprotein (a) was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | 0.0 (8.65) | -27.1 (31.19)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance was concluded if p ≤0.05. No further adjustments were made for tertiary parameters

13. Other Pre Specified Outcome: Lipoprotein (a) at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 37.3 (76.3) | 53.5 (45.8)
  Primary efficacy time point | 41.3 (90.1) | 42.3 (48.2)

14. Other Pre Specified Outcome: Percent Change From Baseline in Very Low Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: Very low density lipoprotein cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | 4.6 (26.53) | -27.1 (30.79)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — Statistical significance was concluded if p ≤0.05. No further adjustments were made for tertiary parameters

15. Other Pre Specified Outcome: Very Low Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 29.8 (12.7) | 28.3 (10.2)
  Primary efficacy time point | 29.8 (12.5) | 19.4 (9.5)

16. Other Pre Specified Outcome: Percent Change From Baseline in the Ratio of Low-Density Lipoprotein Cholesterol to High-Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: The ratio of low-density lipoprotein (LDL) cholesterol to high-density lipoprotein (HDL) cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | 1.4 (12.84) | -49.2 (22.16)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance was concluded if p ≤0.05. No further adjustments were made for tertiary parameters

17. Other Pre Specified Outcome: Ratio of Low-Density Lipoprotein Cholesterol to High-Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
ratio
  Baseline | 5.3 (2.18) | 5.2 (2.38)
  Primary efficacy time point | 5.4 (2.27) | 2.7 (2.21)

18. Other Pre Specified Outcome: Percent Change From Baseline in Apolipoprotein A1 at the Primary Efficacy Time Point
Description: Apolipoprotein A1 was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | -1.2 (11.11) | -0.0 (12.45)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.784, t-test, 2 sided — Statistical significance was concluded if p ≤0.05. No further adjustments were made for tertiary parameters

19. Other Pre Specified Outcome: Apolipoprotein A1 at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 150.0 (24.8) | 150.3 (25.6)
  Primary efficacy time point | 148.9 (33.2) | 149.1 (24.0)

20. Other Pre Specified Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: High-density lipoprotein cholesterol (HDL-C) was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
percentage of baseline | -2.3 (12.72) | 8.1 (17.15)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.079, t-test, 2 sided — Statistical significance was concluded if p ≤0.05. No further adjustments were made for tertiary parameters

21. Other Pre Specified Outcome: High-Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 12 | 21
mg/dL
  Baseline | 48.8 (12.4) | 48.8 (9.9)
  Primary efficacy time point | 48.5 (16.9) | 52.4 (12.4)

ADVERSE EVENTS:
Time Frame: Day 1 to week 28. On-treatment AEs started on/after the first study drug dose and on/before the end of the treatment period. The treatment period was the time study drug was administered until the later of the PET or 14 days after last study drug dose.
Description: The Safety Set includes all randomized patients who receive at least 1 injection of the study treatment. In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Placebo | Mipomersen
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/21
Other Adverse Events (participants affected / at risk) | 12/12 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Mipomersen (N=21)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Mipomersen (N=21)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Eye allergy (Eye disorders) | 0 | 1
Eye inflammation (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Panophthalmitis (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 2
Faeces hard (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Intestinal functional disorder (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 6
Tooth disorder (Gastrointestinal disorders) | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 8
Feeling abnormal (General disorders) | 1 | 1
Feeling cold (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Influenza like illness (General disorders) | 6 | 10
Injection site discolouration (General disorders) | 0 | 13
Injection site discomfort (General disorders) | 1 | 6
Injection site erythema (General disorders) | 0 | 18
Injection site exfoliation (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 7 | 12
Injection site induration (General disorders) | 1 | 11
Injection site inflammation (General disorders) | 0 | 4
Injection site nodule (General disorders) | 0 | 3
Injection site pain (General disorders) | 2 | 14
Injection site pallor (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 0 | 10
Injection site reaction (General disorders) | 0 | 2
Injection site swelling (General disorders) | 0 | 9
Injection site vesicles (General disorders) | 0 | 1
Injection site warmth (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Sensation of pressure (General disorders) | 1 | 0
Tenderness (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 2
Vessel puncture site reaction (General disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 11
Eye infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 3 | 1
Injection site cellulitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 8
Oral herpes (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time (Investigations) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 6
Albumin urine present (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood phosphorus decreased (Investigations) | 1 | 2
Blood potassium increased (Investigations) | 1 | 0
Body temperature decreased (Investigations) | 0 | 3
Body temperature increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1
Coagulation test abnormal (Investigations) | 0 | 1
Electrocardiogram poor R-wave progression (Investigations) | 0 | 1
Gastric pH decreased (Investigations) | 0 | 1
Globulins decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Protein urine present (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Sputum abnormal (Investigations) | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 9
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Aphonia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 3
Dizziness postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 9
Migraine with aura (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 2
Poor quality sleep (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Listless (Psychiatric disorders) | 0 | 2
Tension (Psychiatric disorders) | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 0 | 2
Vasodilatation (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution will submit for review a proposed publication or presentation at least 90 days prior to submission date. Sponsor has the right to delay publication or presentation for not more than 6 months to address patent applications. Sponsor also has the right to demand in writing the deletion of confidential information. Investigator will not make public raw study data, detailed subject cases, or information identifying any subject.